CLINICAL TRIAL: NCT03248869
Title: Asthma Mobile Health Application 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Apple Inc. (Industry); Lifemap Solutions, Inc (Unknown); Sage Bionetworks (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: GCO 15-0063
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: asthma; mobile application; mobile app; mobile health applications; asthma mobile health application
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: A/B testing is a randomized statistical experiment with intervention and control study arms, A and B. New users, as of December 2015, will be stratified and randomized to different daily survey formats in order to test differences in daily survey participation rates. Since this was a mobile "app" based study, a first of its kind - which was available in the App store, it was possible to recruit widely in large numbers. Therefore, even though this was a feasibility study, the sample size was large.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current Daily Survey (Active Comparator): need description
  Interventions: Other: Current Daily Survey
- Mobile Health App (MHA) (Experimental): Participants download the mobile health app via the Apple App Store
  Interventions: Other: Mobile Health App

INTERVENTIONS:
Other: Current Daily Survey — need description
  Arms: Current Daily Survey
Other: Mobile Health App — Participants recruited, consented and enrolled via the AMHA and complete assessments using the app
  Other Names: Asthma Mobile Health App
  Arms: Mobile Health App (MHA)

SUMMARY:
Mobile health applications (MHA) are increasingly being explored as tools to assist in management of chronic diseases. Little is known regarding which characteristics of MHAs are effective and there is limited data suggesting a real-world impact on health outcomes. Asthma is one of the most common and costly of the chronic diseases, impacting a broad range of the population including both children and adults. It is a variable disease necessitating regular medication use, monitoring of symptoms, and avoidance of specific triggers. These characteristics of asthma make it a chronic disease that is particularly amenable to having an MHA facilitate active monitoring outside of periodic traditional medical visits. The study team has designed a MHA focused on asthma subjects to test the feasibility of an asthma mobile health application (AMHA). The AMHA 2.0 study is the result of a collaboration between MHA developers and Mount Sinai faculty with expertise in the fields of asthma, research design, data storage, and data analysis. AMHA 2.0 incorporated elements of usual clinical care (that may take place during typical office visits), such as medication reminders, a daily asthma diary to track asthma control (AC) and medication use, patient education and assessments of quality of life (QoL), and health care utilization (HCU).

DETAILED DESCRIPTION:
Mobile health applications (MHA) are increasingly being explored as tools to assist in management of chronic diseases. Little is known regarding which characteristics of MHAs are effective and there is limited data suggesting a real-world impact on health outcomes. Asthma is one of the most common and costly of the chronic diseases, impacting a broad range of the population including both children and adults. It is a variable disease necessitating regular medication use, monitoring of symptoms, and avoidance of specific triggers. These characteristics of asthma make it a chronic disease that is particularly amenable to having an MHA facilitate active monitoring outside of periodic traditional medical visits. The study team has designed a MHA focused on asthma subjects to test the feasibility of an asthma mobile health application (AMHA). The AMHA 2.0 study is the result of a collaboration between MHA developers and Mount Sinai faculty with expertise in the fields of asthma, research design, data storage, and data analysis. AMHA 2.0 incorporated elements of usual clinical care (that may take place during typical office visits), such as medication reminders, a daily asthma diary to track asthma control (AC) and medication use, patient education and assessments of quality of life (QoL), and health care utilization (HCU).

During the AMHA 2.0 study, the aims are to evaluate the feasibility of:

1. Consenting and enrolling a small cohort of subjects with asthma recruited from Mount Sinai pulmonary clinics remotely via downloading the app
2. Feasibility of use of an asthma e-diary and automated e-reminders for medications in this small cohort for one month
3. Exploring if a small cohort of participants will share data from wearable health and fitness monitoring devices if they own and use such devices.

The primary enrollment period for AMHA 2.0 was met in September 2015. More than 7,000 individuals e-consented for the AMHA 2.0 study, providing more than 80,000 survey responses with many participants granting AMHA 2.0 investigators access to geo-location and wellness data. Data collected during the first six months of the AMHA 2.0 study has provided evidence to answer all primary outcome measures.

Continuation of the AMHA 2.0 protocol was approved in December 2015, expanding the study to a larger population who will be followed for a more extended period of time and will be recruited via availability of the AMHA in the Apple App Store in the US, UK, and Ireland. The latest modification submitted in January, adds an entirely new aim, OM6 and SA6, to the project to include a genetics module. The objectives for the continuation study are:

1. To determine the feasibility of recruiting, consenting and enrolling a larger number of subjects remotely via the Apple App Store without direct participant contact during any phase of the study
2. Assess the impact of continued use of an asthma e-diary and automated medication e-reminders for up to 2 years
3. Explore the feasibility of sharing of data from wearable health and fitness monitoring devices (if applicable) from a larger cohort of patients for up to 2 years
4. To test the medical accuracy of algorithms that may be used in future app versions to give specific feedback to participants based on information they input into the AMHA
5. To investigate the association between DNA variants and asthma phenotypes including: asthma severity, symptom patterns, and medication use/response

This second phase of research is designed to continue the process of developing an AMHA that facilitates asthma self-monitoring, promotes positive behavioral changes, and reinforces adherence to treatment plans according to current asthma guidelines, all in a user-friendly fashion conducive to long term use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Self-reported physician diagnosed asthma
* Have an iPhone
* Sufficient English-language ability to participate in informed consent process, complete study assessments and understand the text in mobile phone-delivered interventions

Exclusion Criteria:

* <18 years of age
* Not currently taking any asthma medications
* Does not own an iPhone or know how to handle a mobile phone
* Are unable to read or understand the study materials
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7752 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Number of downloads | 2 years
  Number of people who downloaded AMHA
Percent of participants who aborted study participation | 2 years
  Percent of aborted study participants before completion inclusion/exclusion criteria

SECONDARY OUTCOMES:
Frequency of use of the Daily asthma diary | 2 years
  Feasibility and implied participant acceptability by counting frequency of use of app
Frequency of use of the Asthma Control (AC) questionnaire | 2 years
  Feasibility and implied participant acceptability by counting frequency of use of app
Frequency of use of the Health Care Utilization (HCU) questionnaire | 2 years
  Feasibility and implied participant acceptability by counting frequency of use of app
Percent of completion of Daily asthma diary | 2 years
  Feasibility and implied participant acceptability by counting percent of completion of features in AMHA
Percent of completion of the Asthma Control (AC) questionnaire | 2 years
  Feasibility and implied participant acceptability by counting percent of completion of features in AMHA
Percent of completion of the Health Care Utilization (HCU) questionnaire | 2 years
  Feasibility and implied participant acceptability by counting percent of completion of features in AMHA
Frequency of use of optional AMHA features | 2 years
  Feasibility and implied participant acceptability by frequency of use of optional AMHA features
Asthma Control (AC) questionnaire | up to 6 months
  Daily asthma diary to track asthma control. AC is based o modified GOAL criteria. Total scale range is from 0 (no impairment) 6 (maximal impairment for symptoms and rescue use)
EuroQol 5D-5L (EQ-5D-5L) | up to 6 months
  EuroQol 5D-5L used to measure quality of life: 5 items are scored from 1 (no problems) to 5 (extreme severe problems). The numerals 1-5 have no arithmetic properties and should not be used as a cardinal scale. total of 3125 possible health states is defined in this way. Each state is referred to in terms of a 5 digit code. For example, state 11111 indicates no problems on any of the 5 dimensions, while state 55555 indicates severe problems in each item.
Health Care Utilization (HCU) score | up to 6 months
  Questionnaire regarding HCU events with scores from 0 (no health services used to 10 (all health care service options utilized).
Associations between genetic markers and asthma severity | 2 years
  Statistically significant associations between DNA variants and asthma severity. Clustering, regression, and ensemble statistical models will be employed to partition AMHA 2.0 participants into distinct phenotypic classes.
Associations between genetic markers and symptom patterns | 2 years
  Statistically significant associations between DNA variants and symptom patterns. Clustering, regression, and ensemble statistical models will be employed to partition AMHA 2.0 participants into distinct phenotypic classes.
Associations between genetic markers and medication use/response | 2 years
  Statistically significant associations between DNA variants and medication use/response. Clustering, regression, and ensemble statistical models will be employed to partition AMHA 2.0 participants into distinct phenotypic classes.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-feng Y Chan, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Dept. of Genetics and Genomic Sciences, Icahn Institute for Genomics and Multiscale Biology, Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Murphy KR, Meltzer EO, Blaiss MS, Nathan RA, Stoloff SW, Doherty DE. Asthma management and control in the United States: results of the 2009 Asthma Insight and Management survey. Allergy Asthma Proc. 2012 Jan-Feb;33(1):54-64. doi: 10.2500/aap.2011.32.3518. Epub 2011 Dec 15. PMID 22309716
- [Background] Demoly P, Annunziata K, Gubba E, Adamek L. Repeated cross-sectional survey of patient-reported asthma control in Europe in the past 5 years. Eur Respir Rev. 2012 Mar 1;21(123):66-74. doi: 10.1183/09059180.00008111. PMID 22379176
- [Background] Eakin MN, Rand CS. Improving patient adherence with asthma self-management practices: what works? Ann Allergy Asthma Immunol. 2012 Aug;109(2):90-2. doi: 10.1016/j.anai.2012.06.009. No abstract available. PMID 22840247
- [Background] Tran N, Coffman JM, Sumino K, Cabana MD. Patient reminder systems and asthma medication adherence: a systematic review. J Asthma. 2014 Jun;51(5):536-43. doi: 10.3109/02770903.2014.888572. Epub 2014 Feb 13. PMID 24506699
- [Background] Foster JM, Usherwood T, Smith L, Sawyer SM, Xuan W, Rand CS, Reddel HK. Inhaler reminders improve adherence with controller treatment in primary care patients with asthma. J Allergy Clin Immunol. 2014 Dec;134(6):1260-1268.e3. doi: 10.1016/j.jaci.2014.05.041. Epub 2014 Jul 22. PMID 25062783
- [Background] Marcano Belisario JS, Huckvale K, Greenfield G, Car J, Gunn LH. Smartphone and tablet self management apps for asthma. Cochrane Database Syst Rev. 2013 Nov 27;2013(11):CD010013. doi: 10.1002/14651858.CD010013.pub2. PMID 24282112
- [Background] Bateman ED, Boushey HA, Bousquet J, Busse WW, Clark TJ, Pauwels RA, Pedersen SE; GOAL Investigators Group. Can guideline-defined asthma control be achieved? The Gaining Optimal Asthma ControL study. Am J Respir Crit Care Med. 2004 Oct 15;170(8):836-44. doi: 10.1164/rccm.200401-033OC. Epub 2004 Jul 15. PMID 15256389
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Kumar R, Seibold MA, Aldrich MC, Williams LK, Reiner AP, Colangelo L, Galanter J, Gignoux C, Hu D, Sen S, Choudhry S, Peterson EL, Rodriguez-Santana J, Rodriguez-Cintron W, Nalls MA, Leak TS, O'Meara E, Meibohm B, Kritchevsky SB, Li R, Harris TB, Nickerson DA, Fornage M, Enright P, Ziv E, Smith LJ, Liu K, Burchard EG. Genetic ancestry in lung-function predictions. N Engl J Med. 2010 Jul 22;363(4):321-30. doi: 10.1056/NEJMoa0907897. Epub 2010 Jul 7. PMID 20647190
- [Background] Park HW, Tantisira KG, Weiss ST. Pharmacogenomics in asthma therapy: where are we and where do we go? Annu Rev Pharmacol Toxicol. 2015;55:129-47. doi: 10.1146/annurev-pharmtox-010814-124543. Epub 2014 Sep 29. PMID 25292431
- [Background] Wechsler ME, Kunselman SJ, Chinchilli VM, Bleecker E, Boushey HA, Calhoun WJ, Ameredes BT, Castro M, Craig TJ, Denlinger L, Fahy JV, Jarjour N, Kazani S, Kim S, Kraft M, Lazarus SC, Lemanske RF Jr, Markezich A, Martin RJ, Permaul P, Peters SP, Ramsdell J, Sorkness CA, Sutherland ER, Szefler SJ, Walter MJ, Wasserman SI, Israel E; National Heart, Lung and Blood Institute's Asthma Clinical Research Network. Effect of beta2-adrenergic receptor polymorphism on response to longacting beta2 agonist in asthma (LARGE trial): a genotype-stratified, randomised, placebo-controlled, crossover trial. Lancet. 2009 Nov 21;374(9703):1754-64. doi: 10.1016/S0140-6736(09)61492-6. PMID 19932356
- See also: CDC Vital Signs May 2011, accessed 9/13/14 — https://www.cdc.gov/vitalsigns/
- See also: Global Strategy for Asthma Management and Prevention, Global Initiative for Asthma (GINA) 2014. — http://ginasthma.org